CLINICAL TRIAL: NCT02486978
Title: Effects of Polyphenols Found in Pomegranate and Olives Food Supplements on Postprandial Blood Glucose in Vivo.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Hilda Nyambe, PhD student, University of Leeds
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: MEEC 14-029
Record Dates: First submitted 2015-06-02; First posted 2015-07-01 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Hyperglycaemia
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (no supplement) (Placebo Comparator): Reference will be white bread to give 50 g available carbohydrates with placebo capsule
  Interventions: Other: Control (109 g white bread); Dietary Supplement: Dose 1; Dietary Supplement: Dose 2
- Dose 1 (Experimental): Test will comprise white bread to give 50 g available carbohydrates and one capsule of pomegranate/olive and one capsule placebo
  Interventions: Other: Control (109 g white bread); Dietary Supplement: Dose 1; Dietary Supplement: Dose 2
- Dose 2 (Experimental): Test will comprise white bread to give 50 g available carbohydrates and 2 capsules of pomegranate/olive.
  Interventions: Other: Control (109 g white bread); Dietary Supplement: Dose 1; Dietary Supplement: Dose 2

INTERVENTIONS:
Other: Control (109 g white bread) — Control meal of 109 g white bread to which the response of the test meals with dietary supplements will be compared to.
Dietary Supplement: Dose 1 — The test meal will contain a single dose of the supplements whose response will be compared to that of the control meal.
Dietary Supplement: Dose 2 — The test meal will contain a double dose of the supplements whose response will be compared to that of the control meal.

SUMMARY:
Consumption of carbohydrate containing foods or sugary drinks brings about changes to the blood glucose levels. After a meal or drink, blood glucose rises until it reaches a peak concentration usually after 30 minutes. When the body senses the increase in blood glucose, a hormonal process involving insulin takes place to ensure that the glucose is taken up from the blood for storage and where it is needed for energy in the body. This process then brings about a decrease in the concentration of glucose until it reaches approximately the starting concentration. The original concentration of glucose is attained approximately 2 hours after eating or drinking a carbohydrate food or sugary drink respectively in healthy people.

Different carbohydrates and sugary drinks have different effects on blood glucose response depending on the amount as well as the type of carbohydrate. Those that give rise to a high glucose response compared to a reference carbohydrate (usually glucose) are said to be high glycaemic index (GI) foods and those with a lower glucose response compared to a reference carbohydrate (usually glucose) are said to be low glycaemic index (GI) foods.

Research has shown that diets that give rise to a high glucose response are associated with a number of abnormalities like increased risk of metabolic syndrome. Metabolic syndrome mostly comprises of insulin resistance and glucose intolerance which gives an increased risk of type 2 diabetes. It also gives rise to other conditions like high blood pressure (arterial hypertension), elevated blood insulin levels (hyper-insulinemia), elevated amounts of fat in the liver (fatty hepatosis) and elevated amounts of lipids in the blood (dyslipidemia). After type 2 diabetes become clinically apparent, the risk of cardiovascular disease also rises. Research has also shown that foods/drinks which raise blood glucose levels gradually (low GI) rather than rapidly (high GI) have health benefits which include reducing the risk of metabolic syndrome. Laboratory studies have shown that polyphenols found in fruits, vegetables and plant based foods have a positive effect on carbohydrate metabolism and can lower the blood glucose levels.

This research will determine whether the presence of polyphenols in the diet has any lowering effect on the blood glucose levels and hence the glycaemic index of foods. This will be determined by asking volunteers to consume commercially available food supplements together with white bread and then determining the glycaemic response. The blood glucose response of bread will be determined initially as a control reference. All will be consumed in random order.

Analysis will be done by measuring blood glucose response after consumption of the control reference meal and the test meal containing polyphenols and then determining the incremental area under the glucose curve.

POMEGRANATE AND OLIVE STUDIES WILL BE TREATED SEPARATELY FOR PURPOSES OF PUBLISHING RESULTS. EACH STUDY WILL AIM TO HAVE AT LEAST 16 PARTICIPANTS.

DETAILED DESCRIPTION:
The world health organisation has reported that over 220 million people suffer from diabetes worldwide and that by the year 2030, this number will be doubled. The WHO also reports that in 2004, about 3.4 million people died from high blood sugar. About 90% of all diabetes cases is due to type II diabetes. Type 2 diabetes is largely due to overweight and lack of physical activity characterised by high glucose levels (hyperglycaemia).

In the human diet, the source of blood glucose is carbohydrates. Dietary carbohydrate is important to maintain glycaemic homeostasis and provides the most of the energy in the diets of most people. The control of blood glucose is a hormonal process and it is very important to human physiology. Hormonal processes involve the release of insulin from the β- cells of the pancreatic cells which stimulates the uptake of glucose after a meal, to other tissues either for utilisation (glycolysis) or to be stored in the liver as glycogen (glycogenesis). When blood glucose falls below normal, glucagon is secreted from the pancreatic α-cells and it promotes liver glucose production by inducing the generation of glucose from non-carbohydrate substrates such as amino and fatty acids (gluconeogenesis) and the generation of glucose from glycogen (glycogenolysis).

When the glucose homeostasis hormonal control fails, it entails high blood glucose levels (postprandial hyperglycaemia) which can lead to metabolic syndrome which includes obesity, impaired glucose tolerance (IGT), hypertension and dyslipidemia. Disturbance of glucose homeostasis can also lead to other symptoms such as inflammation and oxidative stress at the whole body level as well as disturbances of the functionality in several organs as well as diabetes . Therefore, as much as carbohydrates are required in the human body as a major source of energy, too much in the diet can have adverse health effects especially the one with high glycaemic effect.

The proposed mechanism adapted from Aston, 2006 of how carbohydrates may affect human health is that when there is a continual presence of high glycaemic index foods in the diet, this gives rise to postprandial glucose rise as well as high insulin demand to act on the high blood glucose levels in the blood. Postprandial glucose rise and high insulin demand may lead to insulin resistance which is the major component of metabolic syndrome. High insulin demand may also lead to β-cell failure which may also result in hyperglycaemia which is also a cause of insulin resistance. Insulin resistance and hyperglycaemia are risk factors for metabolic syndrome and diabetes type 2.

Scientific evidence suggest that postprandial hyperglycaemia in humans has a major role to play in health priorities like type 2 diabetes and blood glucose control. It has been reported that about 90% of all diabetes cases consist of type 2 diabetes. Apart from type I and type 2 diabetes, there are other related conditions which include pre-diabetes (impaired glucose tolerance (IGT) and impaired fasting glucose (IFG) as well as metabolic syndrome (obesity, hypertension and insulin resistance). It has been reported that pre-diabetes and metabolic syndrome increases the risk of developing cardiovascular disease and diabetes mellitus. The glycaemic index was originally proposed with the aim of managing diabetes. However, recent studies have shown that the GI has potential in the prevention of type 2 diabetes as well as in the treatment of metabolic syndrome. Research has shown that high GI diets are associated with increased risk of developing type 2 diabetes . More research has shown that high GI diet is associated with a number of abnormalities like increased metabolic syndrome and insulin resistance. In the same way, a low GI diet is said to improve insulin sensitivity but more research is needed to support this. A few studies have shown this to be the case. However it was observed that it was difficult to know whether this was as a result of improved insulin sensitivity, or improved insulin secretion or due to reduced rate of glucose absorption.

Potential solution Having anything in the diet that can either slow down the digestion and absorption of carbohydrates can help reduce the risk . Among others, two potential solutions are that of consumption of low glycaemic index foods or having ingredients in the diet that can reduce the glycaemic index of foods as well as postprandial blood glucose levels. The presence of inhibiting components in the diet that can reduce postprandial glucose can also be a solution to reducing the risk. Drugs like acarbose are currently used in some countries for the management of type 2 diabetes which act by inhibiting carbohydrate digestive enzymes. However, the use of acarbose has side effects such as nausea, flatulence and diarrhoea. It has been reported that polyphenols also have the potential to inhibit the rise in blood glucose by hindering the rapid absorption of glucose.

A recent review has reported that research using animal models as well as a limited number of human studies, have shown that polyphenols and polyphenol rich foods or beverages have the potential to affect postprandial glycaemic responses and fasting glycaemia as well as an improvement of acute insulin secretion and sensitivity. Other possible mechanisms as reported in the review include pancreatic β- cells stimulation to secrete insulin as well as activation of insulin receptors, modulation of the release of glucose from the liver as well as of intracellular signalling pathways and gene expression.

Another recent review concluded that it is very possible that the effects of polyphenols in the diet will affect glycaemic index of foods as well as postprandial glucose responses in humans. The two mechanisms highlighted by which this can be achieved being the inhibition of sugar metabolising enzymes as well as transporters. This potential action of polyphenols can thus be compared to that of acarbose which acts by the same mechanism and research in chronic intervention studies has shown that it reduces diabetes risk.

This research will involve the use of pomegranate and olive supplements as a source of polyphenols. The study was approved by the University of Leeds Mathematical and Physical Sciences (MAPs) ethical committee with application number MEEC14-029. At least 16 volunteers will be recruited for each supplement (pomegranate or olive). The volunteers will be screened for their fasting blood glucose level. They will need to be healthy and their fasting blood glucose levels should fall within the healthy range of 4.3-5.9mmol/L.

The volunteers are scheduled to attend 3 visits. During each visit, the volunteer comes fasted in the morning and the fasting blood glucose is measured by the use of a glucometer. The volunteer is then given a test meal which will be randomized and blood glucose will be measured at 15, 30, 45, 60, 90, 120,150 and 180 minutes after the first bite of the test meal. The results will be used to plot the area under the curve and results obtained after consuming test meals will be compared to those obtained after consumption of control meals.

POMEGRANATE AND OLIVE STUDIES WILL BE TREATED SEPARATELY FOR PURPOSES OF PUBLISHING RESULTS. EACH STUDY WILL AIM TO HAVE AT LEAST 16 PARTICIPANTS.

ELIGIBILITY:
Inclusion Criteria:

Measured

* Fasting glucose (blood glucose level before breakfast) 3.9 -5.9mmol/L

Self-assessed

* Apparently healthy
* Not diabetic
* Not on long term prescribed medication (except contraceptives)
* Not pregnant or lactating
* Not on special diet (for losing weight or fruit extracts supplements)

Exclusion Criteria:

* Measured
* Fasting glucose (blood glucose level before breakfast) >5.9mmol/L

Self-assessed

* Not healthy
* Diabetic
* On long term prescribed medication (except contraceptives)
* Pregnant or lactating
* On special diet (for losing weight or fruit extracts supplements)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Incremental area under the glucose curve | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gary Williamson, Study Chair — Professor and Chair of Functional foods; Hilda Nyambe, Principal Investigator — Postgraduate research student
Locations (1):
- School of Food Science and Nutrition, Leeds, West Yorkshire, United Kingdom

REFERENCES:
- [Background] Jenkins DJ, Kendall CW, Augustin LS, Franceschi S, Hamidi M, Marchie A, Jenkins AL, Axelsen M. Glycemic index: overview of implications in health and disease. Am J Clin Nutr. 2002 Jul;76(1):266S-73S. doi: 10.1093/ajcn/76/1.266S. PMID 12081850
- [Background] Aston LM. Glycaemic index and metabolic disease risk. Proc Nutr Soc. 2006 Feb;65(1):125-34. doi: 10.1079/pns2005485. PMID 16441952
- [Background] McKeown NM, Meigs JB, Liu S, Saltzman E, Wilson PW, Jacques PF. Carbohydrate nutrition, insulin resistance, and the prevalence of the metabolic syndrome in the Framingham Offspring Cohort. Diabetes Care. 2004 Feb;27(2):538-46. doi: 10.2337/diacare.27.2.538. PMID 14747241
- [Background] Grundy SM, Brewer HB Jr, Cleeman JI, Smith SC Jr, Lenfant C; American Heart Association; National Heart, Lung, and Blood Institute. Definition of metabolic syndrome: Report of the National Heart, Lung, and Blood Institute/American Heart Association conference on scientific issues related to definition. Circulation. 2004 Jan 27;109(3):433-8. doi: 10.1161/01.CIR.0000111245.75752.C6. No abstract available. PMID 14744958
- [Background] Barclay AW, Petocz P, McMillan-Price J, Flood VM, Prvan T, Mitchell P, Brand-Miller JC. Glycemic index, glycemic load, and chronic disease risk--a meta-analysis of observational studies. Am J Clin Nutr. 2008 Mar;87(3):627-37. doi: 10.1093/ajcn/87.3.627. PMID 18326601
- [Background] Hanhineva K, Torronen R, Bondia-Pons I, Pekkinen J, Kolehmainen M, Mykkanen H, Poutanen K. Impact of dietary polyphenols on carbohydrate metabolism. Int J Mol Sci. 2010 Mar 31;11(4):1365-402. doi: 10.3390/ijms11041365. PMID 20480025
- [Derived] Kerimi A, Nyambe-Silavwe H, Gauer JS, Tomas-Barberan FA, Williamson G. Pomegranate juice, but not an extract, confers a lower glycemic response on a high-glycemic index food: randomized, crossover, controlled trials in healthy subjects. Am J Clin Nutr. 2017 Dec;106(6):1384-1393. doi: 10.3945/ajcn.117.161968. Epub 2017 Oct 11. PMID 29021286